CLINICAL TRIAL: NCT05680064
Title: The Effect of Chewing Gum and Exercises of the Tongue, Lip, and Jaw on Salivation, Xerostomia, and Dysphagia in Patients With Sjögren's Syndrome
Brief Title: The Effect of Chewing Gum, Exercises of the Tongue, Lip, Jaw on Salivation, Xerostomia, Dysphagia in Sjögren's Syndrome
Acronym: SS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Vicdan İtişgen, Clinical Nurse Specialist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/92
Record Dates: First submitted 2022-12-04; First posted 2023-01-11 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Sjögren's Syndrome; Xerostomia; Dysphagia; Salivary Flow Rate
Keywords: Xerostomia,Hyposalivation,Mouth Dryness,Sjögren's syndrome
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia; Deglutition Disorders | interventions — SMG1 protein, human

STUDY DESIGN:
Intervention Model Description: experimental research
Masking Description: At the beginning of this study, all participants are informed about in which group they will participate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients who are routinely followed up will be included in the control group. At the end of 15 days, all patients will come to the second interview. The same data collection methods will be repeated after 15 days.
- Gum-Chewing Group (Experimental): In the gum-chewing group, routine follow-up and additional gum-chewing training will be given (at least 10 minutes 4 times a day, preferably before meals and with sugar-free gum). Patients in the Gum Chewing Group will chew gum as recommended for 15 days. At the end of 15 days, all patients will come to the second interview. The same data collection methods will be repeated after 15 days. In the study, the chewing gum group will chew Vivident Xylit Full Fresh Mint Flavored Liquid Filled Sugar-Free Sweetener Gum. The contents of the gum; Sweeteners (Xylitol, Sorbitols, Mannitol, Maltitols, Aspartame, Acesulfame-K), Gum Yeast, Stabilizer (Glycerol), Flavorings, Natural Mint Flavoring, Maltodextrin, Starch, Emulsifiers (E473, Soy Lecithin), Green Tea Extract, Consistency Enhancers (Cellulose Gum, Xanthan Gum), Coconut Oil, Antioxidant (E321), Brightener (Carnauba Wax), Colorant (E133). There is no allergen warning.
  Interventions: Behavioral: Tongue, lip, chin exercise group
- Tongue, lip, chin exercise group (Experimental): In the tongue, lip and chin exercise group, patients who are routinely followed up and who will be given additional tongue, lip and jaw exercises training (at least 10 minutes 4 times a day and preferably before meals) will take place. Patients in Tongue, Lip, Chin Exercise Group will do the tongue, lip and chin exercises as recommended for 15 days. At the end of 15 days, all patients will come the second interview. The same data collection methods are repeated after 15 days. content of the training to be given to the tongue, lip and chin exercise group and the exercise brochure to be given to the patients T.C. Oral-Motor Exercises Brochure published by the Ministry of Health Istanbul Provincial Health Directorate, Basic Evaluation Principles in Treatment Movements book and Specialist. It was determined and prepared in line with the recommendations of physiotherapist İbrahim ÖZDEMİR.
  Interventions: Behavioral: Tongue, lip, chin exercise group

INTERVENTIONS:
Behavioral: Tongue, lip, chin exercise group — In order to evaluate the effect of chewing gum and tongue, lip and chin exercises on salivary flow rate, xerostomia and dysphagia, both intervention groups will work in a determined time frame daily.
  Other Names: gum chewing group
  Arms: Gum-Chewing Group; Tongue, lip, chin exercise group

SUMMARY:
Sjögren's syndrome (SS) is a chronic, systemic and autoimmune disease characterized by inflammation, fibrosis and dysfunction of exocrine glands such as tear and salivary glands. SS is defined as primary SS when it progresses alone without any other rheumatic disease finding, while the definition of secondary SS is used in the presence of another accompanying autoimmune disease. One of the most disturbing symptoms of SS is hyposalivation, xerostomia and dysphagia due to hypofunction of salivary glands. While xerostomia is the patient's subjective perception of dry mouth, hyposalivation is also evaluated objectively by salivary flow rate measurement methods. Studies have reported that 0.9% to 64.8% of patients with SS experience xerostomia and 32% to 72% of them experience dysphagia. It was planned as a randomized controlled study to examine its effect on dysphagia.

DETAILED DESCRIPTION:
Sjögren's syndrome (SS) is a chronic, systemic and autoimmune disease characterized by inflammation, fibrosis, and dysfunction of exocrine glands such as tear and salivary glands. One of the most disturbing symptoms of SS is hyposalivation, xerostomia, and dysphagia due to the hypofunction of salivary glands. While xerostomia is the patient's subjective perception of dry mouth, hyposalivation is also evaluated objectively by salivary flow rate measurement methods (Pinto, 2021). Studies have reported that 0.9% to 64.8% of patients with SS experience xerostomia and 32% to 72% of them experience dysphagia (Orellana et al, 2016).

With the reduction of saliva, patients may experience difficulties in tasting, chewing, swallowing, speaking, and using prosthesis in patients using prostheses (Pinto, 2021). All these negatively affect the quality of life in patients with SS and their treatment is of great importance (Milin et al, 2016; Pinto, 2021). The treatment of dry mouth in patients with SS consists of pharmacological and non-pharmacological stimulation of the salivary glands and the use of artificial saliva preparations (Ramos_casals et al, 2020). Pharmacological methods used in patients with SS have been shown to reduce dry mouth, but these methods are mostly recommended in severe cases (Ramos_casals et al, 2020; Depinoy et al, 2021). In cases where pharmacological methods are not used, non-pharmacological methods such as taste stimulation (lozenge) and mechanical stimulation (gum) are also recommended in the control of dry mouth (Ramos_casals et al., 2020). It is known that chewing gum increases saliva secretion in studies conducted for different patient groups. used in the treatment of xerostomia in patients with SS, but no study has been found examining the relationship between chewing gum and salivation, xerostomia, and dysphagia in patients with SS (Ramos_casals et al, 2020). In the literature review, no study was found in which the effects of the tongue, lip, and jaw exercises on salivation, xerostomia, and dysphagia were evaluated in any patient group. This study was planned to examine the effects of chewing gum and tongue, lip, and jaw exercises on salivation, xerostomia, and dysphagia in patients with SS.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed as SS according to the 2002 American and European Consensus Group SS classification criteria
* Experiencing xerostomia and dysphagia
* Being between the ages of 18-65
* Not using a total denture
* Not having any other serious illness that will cause dry mouth and dysphagia
* Not having difficulty in chewing and tongue, lip, jaw movement
* Have been receiving treatment for SS for at least 3 months
* To be able to continue working physically and mentally

Exclusion Criteria:

* Not wanting to participate in the study
* Wanting to leave work voluntarily

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Simulated and Unsimulated Salivary Flow Rate | At the first interview, stimulated and unstimulated salivary flow rate of the patients will be measured. In the second interview after 15 days, stimulated and unstimulated salivary flow rate will be measured to observe the change in salivary flow rate.
  Unstimulated Salivary Flow Rate: The patient will be placed in the Fawler position. Individuals will be asked to spit into the graduated tube for 5 minutes to collect saliva samples. The amount of saliva accumulated in the tube will be divided by 5 and the amount of saliva per minute (ml/min) will be calculated.
  Stimulated Salivary Flow Rate: The patient will be placed in the fawler position. Warning for collection of saliva samples will be provided with sugar-free gum. Individuals will be asked to hold the gum in their mouth until it becomes soft, chew for a few seconds, and swallow the first saliva formed. Then, they will be asked to continue the chewing movement using both sides of the jaw for 5 minutes and spit the saliva formed into the graduated tube at short intervals. The salivary flow rate will be calculated as ml/min by dividing the amount of saliva obtained after 5 minutes of chewing by the time.

SECONDARY OUTCOMES:
Xerostomia | It will be measured 2 times with a scale, with an interval of 15 days.
  Xerostomia is the patient's subjective perception of dry mouth. The Xerostomia Inventory 11 will be used to evaluate xerostomia. Each item describing the symptoms will be marked between 1 and 5 points according to the degree of severity. The result is an overall score ranging from 11 to 55 points. A higher total score indicates more severe symptoms are present.
Oral health-related quality of life | It will be measured 2 times with a scale, with an interval of 15 days.
  It is the effect of diseases, deficiencies and inadequacies related to oral and dental health on the quality of life. Oral Health Impact Profile will be used. Items will be answered with points between 0 and 4. The lowest possible score is 0, while the highest score is 56. A high total score indicates a poor oral and dental health-related quality of life.
Dysphagia | It will be measured 2 times with a scale, with an interval of 15 days.
  It is a disorder in which swallowing time is prolonged and more force is used to swallow than normal. The Eating Assessment Tool is used to evaluate dysphagia symptom severity and response to treatment. Each item is scored from 0 to 4. The total score ranges from 0 to 40. A score approaching 0 in the questionnaire indicates that the severity of the swallowing disorder decreases, and a score closer to 40 indicates that the severity of the swallowing disorder increases.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma I CINAR, Prof, Principal Investigator — Saglik Bilimleri Universitesi; Muhammet CINAR, Prof, Study Director — Saglik Bilimleri Universitesi; Vicdan ITISGEN, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Vicdan Itişgen, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basakci Calik B, Gur Kabul E, Keskin A, Bozcuk S, Senol H, Cobankara V. Translation and validation of a Turkish version of the Xerostomia Inventory XI in patients with primary Sjogren's syndrome. Turk J Med Sci. 2021 Oct 21;51(5):2477-2484. doi: 10.3906/sag-2005-157. PMID 34165270
- [Background] Başol ME, Karaağaçlıoğlu L, Yılmaz B. Türkçe Ağız Sağlığı Etki Ölçeğinin Geliştirilmesi OHIP-14-TR. Turkiye Klinikleri J Dental Sci. 2014; 20: 85-92.
- [Background] Dalkılıç E, Coşkun BN. Sjögren Sendromunda Sinir Sistemi Tutulumu ve Vaskülit. RAED Dergisi. 2014; 6(2):62-66.
- [Background] Demir N, Serel Arslan S, Inal O, Karaduman AA. Reliability and Validity of the Turkish Eating Assessment Tool (T-EAT-10). Dysphagia. 2016 Oct;31(5):644-9. doi: 10.1007/s00455-016-9723-9. Epub 2016 Jul 12. PMID 27405421
- [Background] Depinoy T, Saraux A, Pers JO, Boisrame S, Cornec D, Marhadour T, Guellec D, Devauchelle-Pensec V, Bressollette L, Jousse-Joulin S. Salivary Glands and Periodontal Changes in a Population of Sjogren's and Sicca Syndrome Treated by Pilocarpine: A Pilot Study. Rheumatol Ther. 2021 Mar;8(1):219-231. doi: 10.1007/s40744-020-00263-y. Epub 2020 Dec 17. PMID 33336287
- [Background] Lopez-Pintor RM, Ramirez L, Serrano J, de Pedro M, Fernandez-Castro M, Casanas E, Hernandez G. Effects of Xerostom(R) products on xerostomia in primary Sjogren's syndrome: A randomized clinical trial. Oral Dis. 2019 Apr;25(3):772-780. doi: 10.1111/odi.13019. Epub 2019 Jan 8. PMID 30561129
- [Background] Milin M, Cornec D, Chastaing M, Griner V, Berrouiguet S, Nowak E, Marhadour T, Saraux A, Devauchelle-Pensec V. Sicca symptoms are associated with similar fatigue, anxiety, depression, and quality-of-life impairments in patients with and without primary Sjogren's syndrome. Joint Bone Spine. 2016 Dec;83(6):681-685. doi: 10.1016/j.jbspin.2015.10.005. Epub 2016 Jan 13. PMID 26774177
- [Background] Mumcu G, Bıçakçıgil M, Cimilli H, Toker, E, Atalay T, Yavuz Ş. Sjögren Sendromlu Hastalarda Ağız Sağlığının Değerlendirilmesi-Pilot Çalışma. EÜ Diş Hek Fak Derg. 2006; 27:39-44.
- [Background] Orellana MF, Lagravere MO, Boychuk DG, Major PW, Flores-Mir C. Prevalence of xerostomia in population-based samples: a systematic review. J Public Health Dent. 2006 Spring;66(2):152-8. doi: 10.1111/j.1752-7325.2006.tb02572.x. PMID 16711637
- [Background] Pinto A. Management of xerostomia and other complications of Sjogren's syndrome. Oral Maxillofac Surg Clin North Am. 2014 Feb;26(1):63-73. doi: 10.1016/j.coms.2013.09.010. PMID 24287194
- [Background] Ramos-Casals M, Brito-Zeron P, Bombardieri S, Bootsma H, De Vita S, Dorner T, Fisher BA, Gottenberg JE, Hernandez-Molina G, Kocher A, Kostov B, Kruize AA, Mandl T, Ng WF, Retamozo S, Seror R, Shoenfeld Y, Siso-Almirall A, Tzioufas AG, Vitali C, Bowman S, Mariette X; EULAR-Sjogren Syndrome Task Force Group. EULAR recommendations for the management of Sjogren's syndrome with topical and systemic therapies. Ann Rheum Dis. 2020 Jan;79(1):3-18. doi: 10.1136/annrheumdis-2019-216114. Epub 2019 Oct 31. PMID 31672775